CLINICAL TRIAL: NCT04902859
Title: Clonidine as Pain Relief During ROP Eye Examinations
Acronym: cloROP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Örebro County (Other)
Collaborators: Uppsala County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 273547
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Retinopathy of Prematurity; Pain, Procedural; Premature Infant Disease
Keywords: retinopathy of prematurity; procedural pain; neonatal
MeSH Terms: conditions — Retinopathy of Prematurity; Pain, Procedural

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: None of the above will be aware of study drug or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Clonidine with eye speculum (Experimental): 4 mcg/kg Clonidine given orally in GI-tube.
  Interventions: Drug: Clonidine Oral Liquid Product
- Placebo with eye speculum (Placebo Comparator): Sterile water corresponding to the same volume as 4 mcg/kg of Clonidine given orally in GI-tube.
  Interventions: Drug: Sterile water
- Clonidine without eye speculum (Experimental): 4 mcg/kg Clonidine given orally in GI-tube.
  Interventions: Drug: Clonidine Oral Liquid Product
- Placebo without eye speculum (Placebo Comparator): Sterile water corresponding to the same volume as 4 mcg/kg of Clonidine given orally in GI-tube.
  Interventions: Drug: Sterile water

INTERVENTIONS:
Drug: Clonidine Oral Liquid Product — Clonidine prepared from pharmacy with 20 mcg/ml concentration.
  Arms: Clonidine with eye speculum; Clonidine without eye speculum
Drug: Sterile water — Sterile water used as placebo
  Arms: Placebo with eye speculum; Placebo without eye speculum

SUMMARY:
Preterm infants are at risk of developing ROP (retinopathy of prematurity), an eye condition that can cause blindness. Preterm infants born before gestation week (GA) 30 are therefor screened regularly with eye examinations. These eye examinations are painful and despite a lot of research no clear method of pain relief have been found. Since pain in the preterm infant can lead to both short- and longterm negative consequences an effective pain relief during these examinations are of importance. In this study we will investigate if Clonidine can be effective as pain-relief during ROP eye examinations.

DETAILED DESCRIPTION:
Infants born before gestational week (GA) 30 who are cared for in neonatal units at the university hospitals in Örebro and Uppsala, Sweden can be included in the study.

According to power calculations 18 infants are needed for a power of 80% and significance level of 0.05 in order to cover for potential dropouts we plan to include 25 infants. Since the eye examinations are performed without eye speculum in Örebro and with eye speculum in Uppsala we plan to include 25 infants at each unit. The patient will be its own control and examined according to the units´ guidelines. Data will be collected during the patients´ first two eye examinations. In order to exclude potential effects of previous pain experience the order of treatment (clonidine/sterile water) will be randomized.

Sixty minutes before the first eye examination the infant will receive Clonidine or sterile water in corresponding volumes in the GI-tube by a nurse. During the examination the infant will be placed on a heated examination table and connected to an oxygen saturation probe (measuring oxygen saturation and heart rate) on one foot and electrodes for Galvanic skin response (GSR) on the other. The ophthalmologist will examine the infants eyes without eye speculum or with eye speculum on the respective unit. The infants face, oxygen saturation and heart rate will be videotaped before, during and after the examination making it possible to perform av PIPP-R pain assessment at a later time.

After the eye examination the ophtalmologist will be asked to estimate hos easy the infant was to examine by putting an "x" somewhere on a 10 centimeter long line where one end signifies "very easy to examine" and the other end signifies "very difficult to examine". The ophtalmologist can also write any other comments regarding the examination on the same form. The same procedure will be repeated during the infants´ second examination, but with the treatment he/she did not receive during the first examination.

ELIGIBILITY:
Inclusion Criteria:

* Infants born before 30 weeks gestation, informed consent from parents

Exclusion Criteria:

* Infants that have received other pain relieving or sedating drugs within 24 hours before the procedure, infants without GI-tube, infants with neurological deficit, infants with known heart arrhythmia, infants with circulatory instability (MAP below GA in weeks)

Ages: 5 Weeks to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PIPP-R | Within 30 sec after procedure started
  Pain assessment scale

SECONDARY OUTCOMES:
GSR | Within 30 sec after procedure started
  Galvanic skin response

CONTACTS AND LOCATIONS:
Locations (1):
- Barn- och Ungdomskliniken, Universitetssjukhuset, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carlsen Misic M, Eriksson M, Normann E, Pettersson M, Blomqvist Y, Olsson E. Clonidine as analgesia during retinopathy of prematurity screening in preterm infants (cloROP): protocol for a randomised controlled trial. BMJ Open. 2022 Sep 22;12(9):e064251. doi: 10.1136/bmjopen-2022-064251. PMID 36137627